CLINICAL TRIAL: NCT05084742
Title: Observational Clinical Trial, Prospective and Multicenter, Measuring the Long-term Performance and Safety of Biodentine™ in Patients Treated for Endodontic Indications
Brief Title: Long-term Performance and Safety of Biodentine™ in Patients Treated for Endodontic Indications
Status: Recruiting | Type: Observational
Sponsor: Septodont (Industry)
Collaborators: EndoData (Unknown); Recherche Clinique en Odontologie (ReCOL) (Network); QualityStat (Unknown)
Responsible Party: Sponsor
Other Study IDs: BIOD2021-03; 2021-A01631-40 (Registry Identifier: French ID-RCB)
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Biodentine™ — Biodentine™ is a bioactive dentin substitute from the " Active Biosilicate Technology® " innovation.
  Study participants were treated from 1 year to 5,5 years ago through an endodontic microsurgery using Biodentine™ used in its endodontic indications, i.e., root end-filling, external or internal root resorption repair, root and furcation perforation repair, apexification, and revitalization procedure by means of revascularization.

SUMMARY:
In this observational, retro-prospective, and multicenter PMCF clinical investigation, Biodentine™, an active dentine substitute for professional dental use only, is evaluated at 10 years post-treatment, in its endodontic indications as followed:

* Repair of root or furcation perforations.
* Repair of root resorptions (internal and external).
* Root-end filling in endodontic surgery (retrograde filling).
* Apexification (tooth with open apex).
* Revitalization procedure by means of revascularization.

Evaluation is done through a 10-year post-treatment follow-up with collection of radiographic, clinical examination and safety data.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, adult or child with permanent study tooth (immature or mature)
* Study tooth treated with an endodontic microsurgery using Biodentine™: all microsurgery including root end-filling, external or internal root resorption repair, root and furcation perforation repair and apexification
* Study tooth treated at least 1 year and no more than 5.5 years before inclusion visit
* Availability of baseline radiographic image of the study tooth
* Patient affiliated to national health insurance
* Patient informed about the study and who confirms his/her consent to participate to the study

Exclusion Criteria:

* Patient treated with anti-cancer therapy in the 5 years prior to the treatment
* Uncontrolled systemic disease 1 month prior to the treatment
* Development of a cancer or a systemic disease just after the treatment
* Participation to an interventional clinical trial at the time of the treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 160 patients with a permanent tooth treated at least 1 year and no more than 5.5 years ago through an endodontic microsurgery using Biodentine™, all microsurgery including root end-filling, external or internal root resorption repair, root and furcation perforation repair, apexification, and revitalization procedure by means of revascularization.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographic success of treatment | At 10 years post-treatment
  The proportion of patients with successfull treatment at 10 years post-surgery will be determined on clinical and radiographic success evidences for each endodontic indication of Biodentine™:
  * In root end-filling
  * In root resorption repair (internal, external)
  * In root and furcation perforation repair
  * In apexification
  * In revitalization procedure by means of revascularization

SECONDARY OUTCOMES:
Number of Adverse Events (AE) and device deficiencies | From treatment onset to 10 years post-treatment
  Safety at 10 years post-surgery will be determined based on the cumulative numbers of Adverse Events (AE) and device deficiencies observed from treatment onset to 10 years post-treatment, for each endodontic indication of Biodentine™:
  * In root end-filling
  * In root resorption repair (internal, external)
  * In root and furcation perforation repair
  * In apexification
  * In revitalization procedure by means of revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Grosgogeat, MD, PhD, Study Director — CHU de Lyon, France; Marie Georgelin Gurgel, MD, Principal Investigator — CHU de Toulouse, France; Anne-Margaux Collignon, MD, Principal Investigator — AP-HP, Hôpital Louis Mourier, Colombes, France; Alexis Gaudin, MD, Principal Investigator — CHU de Nantes, France; Cyril Villat, MD, PhD, Principal Investigator — HCL de Lyon, France; Marie-Paule Gellé, MD, Principal Investigator — CHU de Reims, France; Sandrine Dahan, MD, Principal Investigator — Private dental practice, Paris, France; Grégory Caron, MD, Principal Investigator — Private dental practice, Paris, France; Cauris Couvrechel, MD, Principal Investigator — Private dental practice, Paris, France
Locations (6):
- France (6):
  - AP-HP, Hôpital Louis Mourier, Colombes
  - HCL de Lyon, Lyon
  - CHU de Nantes, Nantes
  - Private dental care office, Paris
  - CHU de Reims, Reims
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No